CLINICAL TRIAL: NCT01756482
Title: Phase 2a Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of GS-5806 in Healthy Volunteers Infected With Respiratory Syncytial Virus (RSV-A Memphis 37b Strain)
Brief Title: Safety and Efficacy Study of GS-5806 in Healthy Volunteers Infected With Respiratory Syncytial Virus (RSV)
Acronym: Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-218-0103
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory; Syncytial; Virus; Infections; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases; Infections | interventions — presatovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GS-5806 (Experimental): GS-5806, powder for oral solution
  Interventions: Drug: GS-5806
- Sugar powder for oral solution in juice (Placebo Comparator): Sugar powder for oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-5806 — GS-5806, powder for oral solution
  Arms: GS-5806
Drug: Placebo
  Arms: Sugar powder for oral solution in juice

SUMMARY:
This study is to evaluate the antiviral effect of GS-5806 in healthy adults infected with a strain of Respiratory Syncytial Virus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Between 18 to 45 years old
* Body Mass Index of 18 to 33 kg/m2

Exclusion Criteria:

* Acute or chronic medical illness
* Positive for Human Immunodeficiency Virus, Hepatitis B or C
* Nose or nasopharynx abnormalities
* Abnormal lung function

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in viral load measurements. | Post initial dose of GS-5806/placebo to Day 12
  Area under the curve for viral load as measured by qRT-PCR assay from the first viral load measurement post initial dose of GS-5806 or placebo through day 12.

SECONDARY OUTCOMES:
Change of baseline symptoms | Innoculation through Day 12
  Change of baseline symptoms post initial dose of GS-5806 or placebo through Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Adeyi Adeyemi, MD, Principal Investigator — Retroscreen Virology
Locations (1):
- Retroscreen Virology, London, United Kingdom

REFERENCES:
- [Derived] DeVincenzo JP, Whitley RJ, Mackman RL, Scaglioni-Weinlich C, Harrison L, Farrell E, McBride S, Lambkin-Williams R, Jordan R, Xin Y, Ramanathan S, O'Riordan T, Lewis SA, Li X, Toback SL, Lin SL, Chien JW. Oral GS-5806 activity in a respiratory syncytial virus challenge study. N Engl J Med. 2014 Aug 21;371(8):711-22. doi: 10.1056/NEJMoa1401184. PMID 25140957